CLINICAL TRIAL: NCT02059499
Title: A Randomized, Phase III Study of Intra-anal Imiquimod 2.5% vs. Topical 5-fluorouracil 5% vs. Observation for the Treatment of High-grade Anal Squamous Intraepithelial Lesions in HIV-infected Men and Women
Brief Title: Imiquimod, Fluorouracil, or Observation in Treating HIV-Positive Patients With High-Grade Anal Squamous Skin Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AMC-088; NCI-2013-02288 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-088 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-088 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2025-05-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anal Intraepithelial Neoplasia; High-grade Squamous Intraepithelial Lesion; HIV Infection
MeSH Terms: conditions — Squamous Intraepithelial Lesions; HIV Infections | interventions — Imiquimod; Fluorouracil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (imiquimod) (Experimental): Patients apply imiquimod intra-anally QD for 16 weeks.
  Interventions: Drug: imiquimod; Other: questionnaire administration; Other: laboratory biomarker analysis
- Arm B (fluorouracil) (Experimental): Patients apply fluorouracil intra-anally BID on days 1-5. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluorouracil; Other: questionnaire administration; Other: laboratory biomarker analysis
- Arm C (observation) (No Intervention): Patients receive no treatment. Patients who still have HSIL at week 20 and who agree to randomization may cross-over to Arm A or B.

INTERVENTIONS:
Drug: imiquimod — Given intra-anally
  Other Names: Aldara; IMQ; R 837
  Arms: Arm A (imiquimod)
Drug: fluorouracil — Given intra-anally
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm B (fluorouracil)
Other: questionnaire administration — Ancillary studies
  Arms: Arm A (imiquimod); Arm B (fluorouracil)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm A (imiquimod); Arm B (fluorouracil)

SUMMARY:
This randomized phase III trial studies imiquimod or fluorouracil to see how well they work compared to observation in treating patients with high-grade anal squamous skin lesions who are human immunodeficiency virus (HIV)-positive. Biological therapies, such as imiquimod, may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether imiquimod or fluorouracil is more effective than observation in treating high-grade anal squamous skin lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of intra-anal imiquimod 2.5% for treatment of anal high-grade squamous intraepithelial lesions (HSIL) compared to observation only.

II. To assess the efficacy of intra-anal topical 5-fluorouracil (fluorouracil) 5% for treatment of anal HSIL compared to observation only.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of intra-anal imiquimod 2.5% and topical 5-fluorouracil 5%.

II. To compare the efficacy of intra-anal imiquimod 2.5% and topical 5-fluorouracil 5%.

III. To assess for partial response of intra-anal imiquimod 2.5% or topical 5-fluorouracil 5% as compared to observation only.

IV. To evaluate the effect of intra-anal imiquimod 2.5% and topical 5-fluorouracil 5% on human papilloma virus (HPV) persistence.

V. To evaluate anal HSIL outcomes at week 44. VI. To evaluate the effect of behavioral patterns including tobacco smoking and sexual activity on treatment efficacy, tolerability and HPV.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Patients apply imiquimod intra-anally once daily (QD) for 16 weeks. (closed as of protocol version 5.0)

ARM B: Patients apply fluorouracil intra-anally twice daily (BID) on days 1-5. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive no treatment. Patients who still have HSIL at week 20 and who agree to randomization may cross-over to Arm A or B.

After completion of study treatment, patients are followed up at weeks 20, 24, 26, 32, 40, and 44.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive; documentation of HIV infection must be based on a federally approved, licensed HIV test performed in conjunction with screening (enzyme linked immunosorbent assay [ELISA], western blot, or other test); alternatively, this documentation may include a record that another physician has documented that the patient has HIV based on prior ELISA and western blot; an approved antibody test will be used to confirm diagnosis; if the physician is treating a patient with combination antiretroviral therapy (cART) with a history of HIV positivity based on an approved antibody test then repeat antibody confirmation is not necessary
* Biopsy-proven HSIL (anal intraepithelial neoplasia 2 (AIN2) and/or AIN3) of the anal canal at either the squamocolumnar junction or distal anus, documented within 60 days prior to enrollment, but not less than 1 week prior to enrollment
* HSIL occupies at least 25% of the circumference of the anal canal at either the squamocolumnar junction or distal anus on high-resolution anoscopy (HRA) at screening or entry based on available biopsy results and visual appearance
* Anal HSIL lesions are visible at study entry and no lesions are suspicious for invasive cancer
* Ability to understand and willing to provide informed consent
* Participants must, in the opinion of the Investigator, be capable of complying with the requirements of this protocol including self-administration of study treatment
* Karnofsky performance status of >= 70%
* Cluster of differentiation (CD)4 count >= 200 within 120 days prior to enrollment or plasma HIV-1 ribonucleic acid (RNA) < 200 copies/mL within 120 days prior to enrollment
* For females, cervical cytology (if having a cervix) and gynecologic evaluation within 12 months prior to enrollment
* Absolute neutrophil count (ANC) > 750 cells/mm^3 within 90 days prior to enrollment
* Hemoglobin >= 9.0 g/dL within 90 days prior to enrollment
* Platelet count >= 75,000/mm^3 within 90 days prior to enrollment

Exclusion Criteria:

* History of anal cancer
* Prior intra-anal use of topical 5-fluorouracil 5% or imiquimod 2.5%, 3.75% or 5% at any point, or use of perianal imiquimod 2.5%, 3.75% or 5% or topical 5-fluorouracil 5% within 6 months prior to enrollment
* Extensive concurrent perianal or lower vulvar HSIL or condyloma requiring a different treatment modality than the study treatment, or treatment that cannot be deferred in observation arm, per examining provider
* Condyloma occupying more than 50% of the circumference of the anal canal or that obscures a satisfactory exam
* Ongoing use of anticoagulant therapy other than aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Acute treatment for an infection (excluding fungal infection of the skin and sexually transmitted infections) or other serious medical illness within 14 days prior to study entry
* Malignancy requiring systemic therapy; note: Kaposi's sarcoma limited to the skin is not exclusionary unless requiring systemic chemotherapy
* Concurrent systemic corticosteroids, cytokines, and immunomodulatory therapy (e.g. interferons)
* Prior history of HPV vaccination
* Treatment for anal or perianal HSIL, low-grade squamous intraepithelial lesion (LSIL) or condyloma within 4 months of entry; please note that infrared coagulation (IRC) or electrocautery of a biopsy site to stop bleeding does not constitute treatment
* Female participants who are pregnant or breastfeeding; women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to initiating study treatment; all women of childbearing potential must be willing to comply with an acceptable birth control regimen to prevent pregnancy while receiving treatment and for 3 months after treatment is discontinued as determined by the Investigator; post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential; (note: a woman of childbearing potential is one who is biologically capable of becoming pregnant; this includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilkin, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (13):
- United States (12):
  - UCLA CARE Center, Los Angeles, California
  - UCSF-Mount Zion, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Louisiana State University Health Sciences Center - New Orleans, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Laser Surgery Care, New York, New York
  - Cornell Clinical Trials Unit, New York Presbyterian Hospital, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pedersen TB, Pachler FR, Rosenberg J, Andresen K. Interventions for anal canal intraepithelial neoplasia. Cochrane Database Syst Rev. 2025 Aug 13;8(8):CD009244. doi: 10.1002/14651858.CD009244.pub3. PMID 40801169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened between December 2015 to August 2022 at one of the 11 AMC sites certified by the HPV Working Group in HRA. Participants were selected from established HSIL-positive clinic patients or referrals from physicians, such as primary care physicians, HIV specialists, dermatologists, or colorectal surgeons.
Pre-assignment Details: 142 patients were screened using HRA, clinical examination and laboratory tests (within 90 days) to ensure they meet the eligibility criteria. 91 patients were considered eligible and assigned to one of the three study arms.
Groups:
- Arm B (5-fluorouracil): Patients apply topical 5-fluorouracil (5-FU) intra-anally BID on days 1-5. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given intra-anally
  questionnaire administration: Ancillary studies
  laboratory biomarker analysis: Correlative studies
Period: Upto Week 20
Arm/Group | Arm A (Imiquimod) | Arm B (5-fluorouracil) | Arm C (Observation)
Started | 18 | 36 | 37
Population for Primary Endpoint (Week 20 Visit) | 18 | 36 | 37
Completed | 15 | 27 | 32
Not Completed | 3 | 9 | 5
Not completed — Lost to Follow-up | 2 | 6 | 0
Not completed — Treatment completed per protocol criteria | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — No treatment per protocol criteria | 0 | 0 | 5
Period: Post-week 20
Arm/Group | Arm A (Imiquimod) | Arm B (5-fluorouracil) | Arm C (Observation)
Started | 15 | 27 | 13 (13 patients continued in observation arm. The remaining 19 patients in Arm C were re-randomized to either 5-FU or imiquimod therapy (details in next table))
Patients Continuing Originally Assigned Treatment | 15 | 27 | 13
Completed | 12 | 20 | 4
Not Completed | 3 | 7 | 9
Not completed — Treatment not as per protocol criteria | 3 | 4 | 9
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Cross-over Post-week 20 (Re-randomized)
Arm/Group | Arm A (Imiquimod) | Arm B (5-fluorouracil) | Arm C (Observation)
Started (This table provides a patient flow for the 19 patients from Arm C, that were re-randomized to 5-FU or Imiquimod therapy at week 20.) | 5 (Patients in arm C randomized to topical imiquimod intra-anal therapy with similar treatment as per arm A) | 14 (Patients in arm C randomized to topical 5-FU intra-anal therapy with similar treatment as per arm B) | 0
Week 44 Visit for Initial Observation Arm Participants Who Crossed Over or Declined Crossover | 5 | 14 | 0
Completed | 5 | 11 | 0
Not Completed | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population, which consists of all participants who were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil) | Arm C (Observation) | Total
Number analyzed (Participants) | 18 | 36 | 37 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (14.3) | 43.1 (12.9) | 44.7 (14.0) | 44.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 13
  Male | 16 | 30 | 32 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 13 | 30
  Not Hispanic or Latino | 14 | 21 | 22 | 57
  Unknown or Not Reported | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 11 | 14 | 30
  White | 9 | 16 | 16 | 41
  More than one race | 1 | 2 | 3 | 6
  Unknown or Not Reported | 2 | 6 | 3 | 11
Cytology at baseline [Count of Participants; unit: Participants]
  Normal | 1 | 1 | 2 | 4
  Atypical Squamous Cells of Undetermined Significance (ASCUS) | 7 | 11 | 12 | 30
  Low-grade Squamous Intraepithelial Lesion (LSIL) | 2 | 3 | 4 | 9
  Atypical Squamous Cells, cannot exclude High-grade Squamous Intraepithelial Lesion (ASC-H) or HSIL | 8 | 21 | 19 | 48
Number of octants involved as per visual appearance and biopsy performed through HRA [Median (Inter-Quartile Range); unit: octant] — Anal canal is divided in either anatomical sections, referred as octants. High-resolution anoscopy (HRA) examination at screening will be performed to assess the extent of HSIL in terms of number of octants involved and will be based on visual appearance and biopsy.
  octant | 4 [3 to 6] | 4 [3 to 6] | 4 [2 to 5] | 4 [3 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response in 5-FU Arm and Observation Arm Using ITT Population
Description: Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology.
  The percentage of participants achieving complete response in the 5-FU and observation arms will be reported and compared across sites, along with the corresponding p-value, using stratified Mantel-Haenszel-Cochran tests at a one-sided alpha level of 0.025.
Time Frame: At week 20
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm C (Observation) | Arm B (Fluorouracil)
Number analyzed (Participants) | 37 | 36
Participants | 5 | 9
Statistical Analysis 1: Comparison: Arm C (Observation) vs Arm B (Fluorouracil); Test type: Superiority; p = 0.1877, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

2. Primary Outcome: Percentage of Participants Achieving Complete Response (5-FU vs Observation ) Using Per Protocol Population
Description: Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology.
  The percentage of participants achieving complete response in the 5-FU and observation arms will be reported, along with the corresponding p-value, using stratified Mantel-Haenszel-Cochran tests to compare results across sites at a one-sided alpha level of 0.025.
Time Frame: At week 20
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 27 | 31
Participants | 9 | 5
Statistical Analysis 1: Comparison: Arm B (Fluorouracil) vs Arm C (Observation); Test type: Superiority; p = 0.1068, Cochran-Mantel-Haenszel — A priori threshold for statistical significance was p=0.05

3. Primary Outcome: Percentage of Participants Achieving Complete Response in 5-FU vs. Imiquimod, Using the ITT Population Restricted to Those Randomized to Either Treatment Prior to the Closure of the Imiquimod Arm.
Description: Complete response is defined as an absence of HSIL histology for all biopsies and the absence of HSIL cytology.
  Compare the percentage of complete response in 5-FU vs Imiquimod arms across sites using stratified CMH test at one-sided 0.05 alpha.
Time Frame: Week 20
Population: ITT population. Since the imiquimod arm was stopped early, this comparison uses only the ITT subset with participants randomized to imiquimod and 5-FU prior to closure of the imiquimod arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil)
Number analyzed (Participants) | 18 | 18
Participants | 5 | 5
Statistical Analysis 1: Comparison: Arm A (Imiquimod) vs Arm B (Fluorouracil); Test type: Superiority; p = 0.8071, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

4. Primary Outcome: Percentage of Participants Achieving Complete Response in 5-FU vs. Imiquimod, Using the PP Population Restricted to Those Randomized to Either Treatment Prior to the Closure of the Imiquimod Arm.
Description: Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology.
  Compare the complete response by 5-FU vs Imiquimod across sites using stratified CMH test at one-sided 0.05 alpha using only the participants randomized to imiquimod and 5-FU prior to closure of the imiquimod arm.
Time Frame: Week 20
Population: PP population restricted to those randomized to either treatment prior to the closure of the imiquimod
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil)
Number analyzed (Participants) | 15 | 14
Participants | 5 | 5
Statistical Analysis 1: Comparison: Arm A (Imiquimod) vs Arm B (Fluorouracil); Test type: Superiority; p = 0.6562, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

5. Primary Outcome: Percentage of Participants Achieving Complete Response in Imiquimod vs Observation Arm, Using ITT Population Restricted to Those Randomized to Either Treatment Prior to the Closure of the Imiquimod Arm.
Description: Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology.
  Compare the complete response by Observation vs Imiquimod across sites using stratified CMH test at two-sided 0.05 alpha using only the participants randomized to imiquimod and observation prior to closure of the imiquimod arm.
Time Frame: Week 20
Population: ITT population restricted to those randomized to either treatment prior to the closure of the imiquimod arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm C (Observation)
Number analyzed (Participants) | 18 | 19
Participants | 5 | 0
Statistical Analysis 1: Comparison: Arm A (Imiquimod) vs Arm C (Observation); Test type: Superiority; p = 0.0141, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

6. Primary Outcome: Percentage of Participants Achieving Complete Response in Imiquimod vs Observation Arm, Using Per Protocol Population Restricted to Those Randomized to Either Treatment Prior to the Closure of the Imiquimod Arm.
Description: as for outcome 5
Time Frame: Week 20
Population: PP population restricted to those randomized to either treatment prior to the closure of the imiquimod arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm C (Observation)
Number analyzed (Participants) | 15 | 18
Participants | 5 | 0
Statistical Analysis 1: Comparison: Arm A (Imiquimod) vs Arm C (Observation); Test type: Superiority; p = 0.0141, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

7. Primary Outcome: Number of Participants With Peri-anal HSIL Confirmed by Histology Across All Study Arms
Description: Perianal HSIL are HSIL lesions detected in peri-anal region; These lesions will be detected by visual inspection using high resolution anoscopy and biopsy.
  Number of participants with presence of peri-anal HSIL on histology
Time Frame: At week 20
Population: Enrolled patients in each study arm
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 18 | 36 | 37
Participants | 1 | 0 | 0

8. Primary Outcome: Number of Participants With Intra-anal HSIL
Description: Intra-anal HSIL lesions are those lesions that are detected in intra-anal region. It will be detected using visual inspection using HRA followed by positive identification of HSIL using biopsy or cytology.
  Presence of intra-anal HSIL lesions will be descriptively reported across the three arms
Time Frame: At week 20
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 18 | 36 | 37
Participants | 12 | 27 | 32

9. Secondary Outcome: Number of Participants Who Experienced an Adverse Event of Grade 1 to 5 by Week 44, Irrespective of Relatedness to the Intervention. AEs Were Stratified According to Those Reported at or Before Week 20 and After Week 20.
Description: Adverse events are graded on a scale from 1 (mild) to 5 (death) as per CTCAE v. 5.0, with higher grades indicating greater severity.
  The number of participants who experienced an adverse event of grade 1 to 5 by Week 44, regardless of its relatedness to the intervention, will be reported.
  AEs were stratified according to those reported at or before Week 20 and after Week 20.
Time Frame: Up to week 44
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Imiquimod)- Up to Week 44: Patients apply imiquimod intra-anally QD for 16 weeks.
  imiquimod: Given intra-anally
  questionnaire administration: Ancillary studies
  laboratory biomarker analysis: Correlative studies
- Arm B (Fluorouracil)- Up to Week 44: Patients apply fluorouracil intra-anally BID on days 1-5. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given intra-anally
  questionnaire administration: Ancillary studies
  laboratory biomarker analysis: Correlative studies
- Arm C (Observation)- Up to Week 20: Patients receive no treatment. Patients who still have HSIL at week 20 and who agree to randomization may cross-over to Arm A or B.
- Arm C (Observation) After Week 20-Imiquimod; Arm C (Observation) After Week 20- Fluorouracil: Participants Initially Randomized to Observation Arm Who Later Crossed Over
- Arm C (Observation) After Week 20-Not Crossed Over: Participants initially randomized to Observation Arm that didn't crossover to either of the treatment arms
Arm/Group | Arm A (Imiquimod)- Up to Week 44 | Arm B (Fluorouracil)- Up to Week 44 | Arm C (Observation)- Up to Week 20 | Arm C (Observation) After Week 20-Imiquimod | Arm C (Observation) After Week 20- Fluorouracil | Arm C (Observation) After Week 20-Not Crossed Over
Number analyzed (Participants) | 18 | 36 | 37 | 5 | 14 | 13
Participants
  Up to week 20: Grade 1 | 0 | 2 | 2 | 0 | 0 | 0
  Up to week 20: Grade 2 | 3 | 4 | 0 | 0 | 0 | 0
  Up to Week 20: Grade 3 | 1 | 2 | 0 | 0 | 0 | 0
  Up to Week 20: Grade 4 | 1 | 1 | 0 | 0 | 0 | 0
  Up to Week 20: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0
  After week 20: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0
  After Week 20: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  After Week 20: Grade 3 | 0 | 2 | 0 | 0 | 1 | 0
  After week 20: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  After Week 20: Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants Achieving Complete or Partial Response in 5-FU vs Observation Using ITT Population
Description: Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology.
  Partial response is defined as either 1) The regression of HSIL histology but HSIL cytology is present, or 2) Reduction in number of octants with HSIL.
  Percentages will be compared across sites using the stratified Mantel-Haenszel-Cochran test at the two-sided 0.05 alpha level.
Time Frame: Up to week 20
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 36 | 37
Participants | 21 | 15
Statistical Analysis 1: Comparison: Arm B (Fluorouracil) vs Arm C (Observation); Test type: Superiority; p = 0.1409, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

11. Secondary Outcome: Percentageof Patients Achieving Complete or Partial Response in Imiquimod vs Observation Arm, Using ITT Population Restricted to Those Randomized to Either Treatment Prior to the Closure of the Imiquimod Arm.
Description: Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology. Partial response is defined as 1) The regression of HSIL histology but HSIL cytology is present, or 2) Reduction in number of octants with HSIL.
  Percentage of patients achieving complete or partial responses with imiquimod will be compared to observation using participants randomized to imiquimod and observation prior to closure of the imiquimod arm.
Time Frame: Up to week 20
Population: ITT population restricted to those randomized to either treatment prior to the closure of the imiquimod arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm C (Observation)
Number analyzed (Participants) | 18 | 19
Participants | 11 | 6
Statistical Analysis 1: Comparison: Arm A (Imiquimod) vs Arm C (Observation); Test type: Superiority; p = 0.0805, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

12. Secondary Outcome: Amount of Drug Consumed in 5-FU and Imiquimod Arm by Week 16
Description: Amount of study drug consumed by measuring the mass of study drug dispensed (weight of study drug container at baseline - weight of study drug at the end of treatment) by study arm (5FU vs imiquimod) by the time of receiving 8 cycle treatment
Time Frame: Week 16
Population: ITT
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil)
Number analyzed (Participants) | 18 | 36
grams | 39.5 (7.7) | 32.6 (17.2)

13. Secondary Outcome: Percentage of Participants Achieving Complete or Partial Response in 5-FU vs Observation Using ITT Population
Description: Complete response is defined as the Complete response is defined as the absence of HSIL histology for all biopsies and the absence of HSIL cytology. Partial response is defined as 1) The regression of HSIL histology but HSIL cytology is present, or 2) Reduction in number of octants with HSIL.
  Percentage will be compared across sites using the stratified Mantel-Haenszel-Cochran test at the two-sided 0.05 alpha level.
Time Frame: At 44 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 36 | 37
Participants | 17 | 19
Statistical Analysis 1: Comparison: Arm B (Fluorouracil) vs Arm C (Observation); Test type: Superiority; p = 0.5726, Cochran-Mantel-Haenszel

14. Secondary Outcome: Percentage of Patients Achieving Complete or Partial Response in Imiquimod vs Observation Arm, Using ITT Population Restricted to Those Randomized to Either Treatment Prior to the Closure of the Imiquimod Arm.
Description: The proportion of patients achieving complete or partial responses with imiquimod will be compared to observation using participants randomized to imiquimod and observation prior to closure of the imiquimod arm. Complete response is defined as the absence of HSIL based on central pathology review, if available; otherwise, local biopsy results will be used. Partial Response is defined as: 1) The regression of HSIL histology but HSIL cytology is present, or 2) Reduction in number of octants with HSIL.
Time Frame: Up to week 44
Population: ITT population restricted to those randomized to either treatment prior to the closure of the imiquimod arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm C (Observation)
Number analyzed (Participants) | 18 | 19
Participants | 11 | 10
Statistical Analysis 1: Comparison: Arm A (Imiquimod) vs Arm C (Observation); Test type: Superiority; p = 0.6184, Cochran-Mantel-Haenszel — The threshold for statistical significance was p=0.05

15. Secondary Outcome: Persistence and New Infections of HPV Type Specific Infections
Description: The proportion of participants with persistent HPV infection, defined as the presence of the same HPV type detected at both baseline and Week 20. The proportion of participants who acquire a new HPV infection at Week 20 that was not detected at baseline is new infection. Persistence and new infection will be assessed separately for each HPV type.
Time Frame: At week 20
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 18 | 36 | 37
Participants
  Persistent : HPV 16 | 1 | 4 | 3
  Persistent : HPV 18 | 1 | 3 | 1
  Persistent : HPV 31 | 1 | 5 | 4
  Persistent : HPV 33 | 0 | 1 | 2
  Persistent : HPV 35 | 0 | 1 | 2
  Persistent : HPV 39 | 0 | 3 | 0
  Persistent : HPV 45 | 0 | 1 | 1
  Persistent : HPV 51 | 1 | 0 | 0
  Persistent : HPV 52 | 0 | 2 | 1
  Persistent : HPV 53 | 1 | 4 | 2
  Persistent : HPV 56 | 1 | 1 | 1
  Persistent : HPV 58 | 2 | 1 | 3
  Persistent : HPV 59 | 0 | 3 | 6
  Persistent : HPV 66 | 0 | 1 | 0
  Persistent : HPV 68 | 2 | 4 | 0
  Persistent: any high-risk HPV infection | 12 | 17 | 25
  New infections : HPV 16 | 5 | 8 | 8
  New infections : HPV 18 | 3 | 1 | 2
  New infections : HPV 31 | 2 | 2 | 5
  New infections : HPV 33 | 3 | 4 | 5
  New infections : HPV 35 | 1 | 3 | 3
  New infections : HPV 39 | 1 | 2 | 2
  New infections : HPV 45 | 2 | 2 | 0
  New infections : HPV 51 | 1 | 3 | 2
  New infections : HPV 52 | 0 | 4 | 4
  New infections : HPV 53 | 2 | 3 | 5
  New infections : HPV 56 | 5 | 5 | 2
  New infections : HPV 58 | 3 | 3 | 3
  New infections : HPV 59 | 3 | 4 | 2
  New infections : HPV 66 | 0 | 2 | 0
  New infections : HPV 68 | 3 | 4 | 3
  New infections: any high-risk HPV | 11 | 21 | 26
  Overall number of patients with hrHPV positivity at week 20 | 12 | 22 | 26

16. Secondary Outcome: Comparison of the Number of hrHPV Genotypes in Each Arm Observed at Baseline vs at Week 20
Description: hrHPV genotypes will be detected in anal swabs specimens processed using polymerase chain reaction (PCR) and reverse line blot analysis.
  Comparison of mean number of hrHPV genotypes in each arm observed at baseline vs at week 20
Time Frame: week 20
Population: Per protocol
Measure: Mean (Standard Deviation); unit: hrHPV genotypes
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 15 | 27 | 31
hrHPV genotypes
  Baseline | 3.75 (1.81) | 4.25 (2.41) | 3.32 (2.01)
  Week 20 | 3.67 (2.06) | 3.5 (2.36) | 2.62 (1.65)
Statistical Analysis 1: Comparison: Arm A (Imiquimod); Comparison of number of hrHPV genotypes in each arm observed at baseline vs at week 20 in imiquimod arm; Test type: Equivalence — Comparison of mean between count of hrHPV genotypes observed at baseline vs at week 20 in imiquimod arm; p = 0.3, Wilcoxon (Mann-Whitney) — A priori threshold for interpreting significance : 0.05
Statistical Analysis 2: Comparison: Arm B (Fluorouracil); Comparison of the count of hrHPV genotypes observed at baseline vs at week 20 in 5FU arm; Test type: Equivalence — Comparison of mean number of hrHPV genotypes observed at baseline vs at week 20 in 5FU arm; p = 0.3, Wilcoxon (Mann-Whitney) — A priori threshold to interpret significance: 0.05
Statistical Analysis 3: Comparison: Arm C (Observation); Comparison of the count of hrHPV genotypes observed at baseline vs at week 20 in observation arm; Test type: Equivalence — Comparison of mean number of hrHPV genotypes observed at baseline vs at week 20 in observation arm; p = 0.26, Wilcoxon (Mann-Whitney) — A priori cutoff of significance: 0.05

17. Secondary Outcome: HPV Genotypes Present at Baseline But no Longer Detected at Week 20
Description: Count of HPV genotypes present at baseline but no longer detected at week 20.
Time Frame: 20 weeks
Population: Per protocol
Measure: Count of Units; unit: Unique HPV genotypes
Units Other Than Participants: Unique HPV genotypes
Arm/Group | Arm A (Imiquimod) | Arm B (Fluorouracil) | Arm C (Observation)
Number analyzed (Participants) | 15 | 27 | 31
Number analyzed (Unique HPV genotypes) | 14 | 15 | 15
Unique HPV genotypes
  Count and percentage of unique HPV genotypes undetected at week 20 | 2 | 0 | 1
  Count and percentage of unique HPV genotypes re-detected at week 20 | 12 | 15 | 14

ADVERSE EVENTS:
Time Frame: Upto 44 Weeks
Groups:
- Arm A (Imiquimod)-Up to 44 Weeks: Patients apply imiquimod intra-anally QD for 16 weeks.
  imiquimod: Given intra-anally
  questionnaire administration: Ancillary studies
  laboratory biomarker analysis: Correlative studies
- Arm B (Fluorouracil)- Up to 44 Weeks: Patients apply fluorouracil intra-anally BID on days 1-5. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given intra-anally
  questionnaire administration: Ancillary studies
  laboratory biomarker analysis: Correlative studies
- Arm C (Observation)-Up to 20 Weeks: Patients receive no treatment. Patients who still have HSIL at week 20 and who agree to randomization may cross-over to Arm A or B.
- Arm C (Observation) After Week 20-Imiquimod; Arm C (Observation) After Week 20-Fluorouracil: Patients initially randomized to Observation but later on agreed to crossover
- Arm C (Observation)- After Week 20, Not Crossed Over: Patients didn't crossover to eithe fluorouracil or Imiquimod
Arm/Group | Arm A (Imiquimod)-Up to 44 Weeks | Arm B (Fluorouracil)- Up to 44 Weeks | Arm C (Observation)-Up to 20 Weeks | Arm C (Observation) After Week 20-Imiquimod | Arm C (Observation) After Week 20-Fluorouracil | Arm C (Observation)- After Week 20, Not Crossed Over
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/36 | 0/37 | 0/5 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/18 | 4/36 | 0/37 | 0/5 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 2/18 | 5/36 | 2/37 | 0/5 | 1/14 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Imiquimod)-Up to 44 Weeks (N=18) | Arm B (Fluorouracil)- Up to 44 Weeks (N=36) | Arm C (Observation)-Up to 20 Weeks (N=37) | Arm C (Observation) After Week 20-Imiquimod (N=5) | Arm C (Observation) After Week 20-Fluorouracil (N=14) | Arm C (Observation)- After Week 20, Not Crossed Over (N=13)
INFECTIONS AND INFESTATIONS (BACTEREMIA) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Imiquimod)-Up to 44 Weeks (N=18) | Arm B (Fluorouracil)- Up to 44 Weeks (N=36) | Arm C (Observation)-Up to 20 Weeks (N=37) | Arm C (Observation) After Week 20-Imiquimod (N=5) | Arm C (Observation) After Week 20-Fluorouracil (N=14) | Arm C (Observation)- After Week 20, Not Crossed Over (N=13)
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL DISORDERS (Anal spasms) (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - (pain) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
SURGICAL AND MEDICAL PROCEDURES - (tooth filling) (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
DIARRHEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
PROCTITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS ( irritation and bleeding) (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
ANORECTAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT02059499/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT02059499/ICF_001.pdf